CLINICAL TRIAL: NCT03760627
Title: Evaluation of A Mindfulness Resiliency Training Program for Refugees Living in Jordan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2000024279
Record Dates: First submitted 2018-11-16; First posted 2018-11-30 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Mental Health Issue (E.G., Depression, Psychosis, Personality Disorder, Substance Abuse); Mental Health Wellness 1; War-Related Trauma
MeSH Terms: conditions — Depression; Psychotic Disorders; Personality Disorders; Substance-Related Disorders; War-Related Injuries

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge cluster randomized trial design. The design involves random and sequential crossover of clusters from control to intervention until all clusters are exposed. The controls from the previous session who were available for the parallel portion of the study, will later become the treatment group while another control group is recruited for them, which in turn will become an intervention group and so forth.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Refugees Mindfulness Resiliency Training (Experimental): The Collateral Repair Project (CRP) will conduct a Mindfulness Resiliency Training Program (MRTP) for refugees residing in Amman, Jordan. A small support group will demonstrate to participants techniques that they can use to self-manage their own stress and trauma.
  Interventions: Behavioral: Refugees Mindfulness Resiliency Training
- Control arm (Placebo Comparator): The control group will receive the training after the study group at 2 months and the control group will then become the study group for the new session. A new group of 20 participants will be recruited who will act as a control for that session. The surveys from the control group will be compared with the study group at 0 and 2 months. Each session will last for two months. The control group will receive the training at the end of the two months. This process will be repeated for a total of nine sessions over a total period of 12 months.
  Interventions: Behavioral: Mindfulness Resiliency Training

INTERVENTIONS:
Behavioral: Refugees Mindfulness Resiliency Training — The intervention consists of meditation, guided imagery, yoga and exercise, biofeedback; self-expression in words, drawings, and movement; and small group support to demonstrate to participants techniques that they can use to self-manage their own stress and trauma.
  Arms: Refugees Mindfulness Resiliency Training
Behavioral: Mindfulness Resiliency Training — The intervention consists of meditation, guided imagery, yoga and exercise, biofeedback; self-expression in words, drawings, and movement; and small group support to demonstrate to participants techniques that they can use to self-manage their own stress and trauma.
  Arms: Control arm

SUMMARY:
To estimate the efficacy of a structured, scalable and replicable psychosocial intervention targeting refugees living in Jordan, Amman who have been forced to flee their homes due to regional conflicts.

DETAILED DESCRIPTION:
The study is designed to examine the effects of the Mindfulness Resiliency Training Program (MRTP) conducted at Collateral Repair Project (CRP) on the resilience of refugees. The study group and the control group will be recruited from refugees currently residing in Amman, Jordan who are participating in the MRTP at CRP, an ongoing program independent of our study.

In order to assess the effect of the MRTP on participant resiliency, the three survey tools described above will be used:

1. the Strength and Difficulties Questionnaire (SDQ) as a measure of the individual's degree of traumatization and
2. the Child and Youth Resiliency Measure (CYRM-12) (for adolescents) or the Adult Resiliency Measure (ARM-12) (for adults) as a measure of resiliency

ELIGIBILITY:
Inclusion Criteria:

* Participants who will be recruited in the study are adult and adolescent (13-19 years) refugees, Syrian and non-Syrians, who are currently residing in Amman, Jordan who will be participating in the MRTP at CRP.

Exclusion Criteria:

* Jordanian refugees residing in Amman, Jordan.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Assess Mindfulness Resiliency Adolescents | 2 months
  In order to assess the effect of the Mindfulness Resiliency Training Program (MRTP) on participant resiliency, the Child and Youth Resiliency Measurement (CYRM-12) 12 question assessment tool for adolescents will be used to measure an increase in scores from baseline.
Assess Mindfulness Resiliency Adolescents | 6 months
  In order to assess the effect of the MRTP on participant resiliency, the CYRM-12 for adolescents will be used to measure an increase in scores from baseline.
Assess Mindfulness Resiliency Adults | 2 months
  In order to assess the effect of the MRTP on participant resiliency, the Adult Resiliency Measurement 12 question assessment tool (ARM-12) will be used to measure an improvement in score from pre-intervention baseline.
Assess Mindfulness Resiliency Adults | 6 months
  In order to assess the effect of the MRTP on participant resiliency, the Adult Resiliency Measurement tool (ARM-12) will be used to measure an improvement in score from pre-intervention baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Saquib Lakhani, MD, Principal Investigator — Yale University; Prachi Syngal, MD, Principal Investigator — Yale University
Locations (1):
- Collateral repair Project, Amman, Jordan